CLINICAL TRIAL: NCT03849196
Title: Simultaneous Combination of Bisacodyl Suppository Agent and 1L Polyethylene Glycol Plus Ascorbic Acid is Not Inferior and Comfortable Regimen Compared With 2L Polyethylene Glycol Plus Ascorbic Acid: A Randomized Controlled Study
Brief Title: Effectiveness of Bisacodyl Suppository Agent for Dose Reduction of Low Dose PEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Eun Ran Kim, Clinical associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-05-100
Record Dates: First submitted 2019-02-16; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Bisacodyl; Suppositories

STUDY DESIGN:
Intervention Model Description: prospective, randomized, and observer-blind study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2L PEG-Asc (Experimental): 2L PEG-Asc for bowel preparation
  Interventions: Drug: 2L PEG-Asc
- 1L PEG-Asc & 'Bisacodyl 10Mg Suppository (Active Comparator): 1L PEG-Asc with 'Bisacodyl 10Mg Suppository for bowel preparation
  Interventions: Drug: Bisacodyl 10Mg Suppository; Drug: 1L PEG-Asc

INTERVENTIONS:
Drug: 2L PEG-Asc — PEG-Asc powder
  Other Names: clicool; coolprep
  Arms: 2L PEG-Asc
Drug: Bisacodyl 10Mg Suppository — bisacodyl 10 mg suppository
  Arms: 1L PEG-Asc & 'Bisacodyl 10Mg Suppository
Drug: 1L PEG-Asc — PEG-Asc powder
  Other Names: clicool; coolprep
  Arms: 1L PEG-Asc & 'Bisacodyl 10Mg Suppository

SUMMARY:
Proper bowel cleansing before colonoscopy is an important factor to increase the detection rate of lesions. Low volume polyethylene glycol (PEG) plus ascorbic (PEG-Asc) has reduced the dosage of previous bowel preparation agent, but it still presents discomfort to patients. The aim of this study was to confirm the efficacy and convenience of volume reduction of PEG-Asc by adding bisacodyl suppository at the same day by compared with conventional 2L PEG-Asc.

DETAILED DESCRIPTION:
Eligibility criteria: outpatients between the ages of 20 and 70 years, who were scheduled for colonoscopy between August 2017 and January 2018

Exclusion criteria: patients with a history of gastrointestinal tract surgery, inflammatory bowel disease, severe active colitis, underlying chronic kidney disease, or pregnancy.

Outcome measures: the Boston Bowel Preparation Scale (BBPS)

ELIGIBILITY:
Inclusion Criteria:

* outpatients who were scheduled for colonoscopy between August 2017 and January 2018

Exclusion Criteria:

* History of gastrointestinal tract surgery
* History of inflammatory bowel disease
* History of severe active colitis
* History of chronic kidney disease
* pregnant woman.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS). | 1 hour
  4-point scoring system (0-3) applied to each of the 3 colon segments (right colon including cecum and ascending colon, transverse colon including transverse colon, hepatic and splenic flexure, left colon including descending colon, sigmoid colon, and rectum)

CONTACTS AND LOCATIONS:
Overall Officials: brian.biochem@gmail.com Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No